CLINICAL TRIAL: NCT05610865
Title: Autologous Adipose Tissue Derived Stromal Vascular Fraction Versus Cultured Adipose Derived Stem Cells for the Treatment of Chronic Diabetic Wounds
Brief Title: Efficacy of Adipose Tissue Derived Stem Cells for the Treatment of Diabetic Foot Ulcers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of the Punjab (Other)
Collaborators: Centre of Excellence in Molecular Biology, University of the Punjab, Lahore (Unknown); Higher Education Commission (Pakistan) (Other); Jinnah Burn and Reconstructive Surgery Centre, Lahore (Other Government)
Responsible Party: Principal Investigator, Azra Mehmood, Associate Professor, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEMB-SC02
Record Dates: First submitted 2022-10-26; First posted 2022-11-09 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer; Diabetes Mellitus; Diabetic Foot; Diabetic Foot Infection; Diabetic Foot Ulcer Neuropathic; Foot Ulcer Due to Type 1 Diabetes Mellitus; Foot Ulcer Due to Type 2 Diabetes Mellitus; Foot Ulcer; Diabetes Complications; Chronic Diabetic Ulcer of Left Foot; Chronic Diabetic Foot Ulcer of Right Foot
Keywords: Stromal vascular fraction (SVF), Adipose derived stem cells (ASCs), Diabetic foot ulcer (DFU), Platelet rich plasma (PRP)
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer; Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control; Standard-of-care management (Active Comparator): Saline dressing will be done as a routine care management.
  Interventions: Other: Control; Standard-of-care management
- Only PRP injection (Experimental): Only PRP will be injected at the wound site.
  Interventions: Biological: Only PRP injection
- PRP + SVF injection (Experimental): SVF pellet mixed with PRP will be injected at the wound site after adjusting number of cells.
  Interventions: Biological: PRP + SVF injection
- PRP + ASCs injection (Experimental): Cultured ASCs mixed with PRP will be injected at the wound site after adjusting number of cells.
  Interventions: Biological: PRP + ASCs injection

INTERVENTIONS:
Other: Control; Standard-of-care management — Patients will undergo conventional wound care management.
  Arms: Control; Standard-of-care management
Biological: Only PRP injection — Only PRP injected / cm2 intradermally at the border zone & inside of wound surface bed.
  Arms: Only PRP injection
Biological: PRP + SVF injection — Uncultured cells (SVF) along PRP were mixed, transferred to 1 cc syringes and injected / cm2 intradermally at the border zone & inside of wound surface bed.
  Arms: PRP + SVF injection
Biological: PRP + ASCs injection — Cultured ASCs along PRP were mixed, transferred to 1 cc syringes and injected / cm2 intradermally at the border zone & inside of wound surface bed.
  Arms: PRP + ASCs injection

SUMMARY:
The aim of this study is to evaluate the therapeutic efficacy of uncultured adipose derived stromal vascular fraction (SVF) and cultured adipose derived stem cells (ASCs) both supplemented with platelet rich plasma (PRP) to treat chronic diabetic foot ulcers. It will increase the pragmatic potential of both types of cells as PRP is rich in survival and chemotactic factors. Moreover, the autologous nature of the proposed study will ensure safety of its use in diabetic patients and will unveil the more effective therapeutic option for treatment of foot ulcer wounds.

DETAILED DESCRIPTION:
Under local or general anesthesia, autologous fat will be harvested by using a manual aspiration or syringe-assisted technique. SVF and ASCs isolation from autologous lipoaspirates will be done by enzymatic digestion method (collagenase Type-1 solution for 45 minutes at 37°C). Cell quality assessment will be done prior to transplantation by trypan blue exclusion assay and total populations and fractions of cells identified by immunocytochemistry / flow cytometry. PRP will be derived by centrifugation from 50-100ml blood collected in anticoagulant carrying bag, from patient at the day of transplantation. The injection volume will depend on the wound area of each patient. 2 million cells/ 0.5 ml PRP will be mixed, transferred to 1 cc syringes and injected / cm2 intradermally at the border zone & inside of wound surface bed.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 Diabetes Mellitus
* Age 20-60 years (Male/Female)
* Body mass index 20-30 kg/m2
* Suitable for liposuction
* Condition or Disease: Diabetic Neuropathy
* Wound Type: Chronic foot ulcer
* Approx. wound area: 2 cm2 - 8 cm2
* Wound Condition should be of Wagner's grade I (Limited to soft tissue)
* Duration of wound persistence: 6-24 Weeks
* Transcutaneous oxygen pressure > 30 mmHg, and an ankle brachial pressure index > 0.5.
* Already following an adequate off-loading method
* Provided signed informed consent

Exclusion Criteria:

* Uncontrolled hyperglycemia (HbAlc > 9%)
* Presence of severe clinical sign of infection
* Inability to tolerate off-loading, and poor prognosis diseases including malignant tumors.
* Serious chronic disease i.e hepatic, heart, renal, pulmonary diseases
* Patients with critical limb ischemia and osteomylitis
* Withdrawal of informed consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Interview and visual inspection of ulcers recovery rate | 3 months
  This will be done in terms of diameter (cm2) of wounds, monitored in both cell transplanted and standard care patients after week interval till 3 months.

SECONDARY OUTCOMES:
Percentages (%) of wound closure rate (with respect to time) will be assessed. | 3 months
  Change in wound size (cm2) will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Azra Mehmood, PhD, Principal Investigator — Center of Excellence in Molecular Biology (CEMB, University of the Punjab, Lahore; Sheikh Riazuddin, PhD, Study Director — Jinnah Burn and Reconstructive Surgery Center (JB&RSC), Lahore
Locations (1):
- Stem Cell Laboratory, Jinnah Burn and Reconstructive Surgery Center (JB&RSC), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shao S, Pan R, Chen Y. Autologous Platelet-Rich Plasma for Diabetic Foot Ulcer. Trends Endocrinol Metab. 2020 Dec;31(12):885-890. doi: 10.1016/j.tem.2020.10.003. Epub 2020 Nov 13. PMID 33199085
- [Background] Nolan GS, Smith OJ, Heavey S, Jell G, Mosahebi A. Histological analysis of fat grafting with platelet-rich plasma for diabetic foot ulcers-A randomised controlled trial. Int Wound J. 2022 Feb;19(2):389-398. doi: 10.1111/iwj.13640. Epub 2021 Jun 24. PMID 34169656
- [Background] Carstens MH, Quintana FJ, Calderwood ST, Sevilla JP, Rios AB, Rivera CM, Calero DW, Zelaya ML, Garcia N, Bertram KA, Rigdon J, Dos-Anjos S, Correa D. Treatment of chronic diabetic foot ulcers with adipose-derived stromal vascular fraction cell injections: Safety and evidence of efficacy at 1 year. Stem Cells Transl Med. 2021 Aug;10(8):1138-1147. doi: 10.1002/sctm.20-0497. Epub 2021 Apr 7. PMID 33826245
- [Background] Qin HL, Zhu XH, Zhang B, Zhou L, Wang WY. Clinical Evaluation of Human Umbilical Cord Mesenchymal Stem Cell Transplantation After Angioplasty for Diabetic Foot. Exp Clin Endocrinol Diabetes. 2016 Sep;124(8):497-503. doi: 10.1055/s-0042-103684. Epub 2016 May 24. PMID 27219884
- [Background] Han SK, Kim HR, Kim WK. The treatment of diabetic foot ulcers with uncultured, processed lipoaspirate cells: a pilot study. Wound Repair Regen. 2010 Jul-Aug;18(4):342-8. doi: 10.1111/j.1524-475X.2010.00593.x. Epub 2010 May 11. PMID 20492632
- [Background] Didangelos T, Koliakos G, Kouzi K, Arsos G, Kotzampassi K, Tziomalos K, Karamanos D, Hatzitolios AI. Accelerated healing of a diabetic foot ulcer using autologous stromal vascular fraction suspended in platelet-rich plasma. Regen Med. 2018 Apr;13(3):277-281. doi: 10.2217/rme-2017-0069. Epub 2018 May 1. PMID 29715071
- [Background] Prakasam N, Prabakar MS, Reshma S, Loganathan K, Senguttuvan K. A clinical study of platelet rich plasma versus conventional dressing in management of diabetic foot ulcers. International Surgery Journal. 2018 Sep 25;5(10):3210-6.
- [Background] Alvaro-Afonso FJ, Sanz-Corbalan I, Lazaro-Martinez JL, Kakagia D, Papanas N. Adipose-Derived Mesenchymal Stem Cells in the Treatment of Diabetic Foot Ulcers: A Review of Preclinical and Clinical Studies. Angiology. 2020 Oct;71(9):853-863. doi: 10.1177/0003319720939467. Epub 2020 Jul 29. PMID 32723090
- [Background] Khan A, Junaid N. Prevalence of diabetic foot syndrome amongst population with type 2 diabetes in Pakistan in primary care settings. J Pak Med Assoc. 2017 Dec;67(12):1818-1824. PMID 29256523
- [Background] Yin S, Yang X, Bi H, Zhao Z. Combined Use of Autologous Stromal Vascular Fraction Cells and Platelet-Rich Plasma for Chronic Ulceration of the Diabetic Lower Limb Improves Wound Healing. Int J Low Extrem Wounds. 2021 Jun;20(2):135-142. doi: 10.1177/1534734620907978. Epub 2020 Mar 4. PMID 32131655